CLINICAL TRIAL: NCT00125788
Title: A Phase II, Prospective, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study of L Glutamine Therapy for Sickle Cell Anemia and Sickle ß0-Thalassemia
Brief Title: L-Glutamine Therapy for Sickle Cell Anemia and Sickle ß0 Thalassemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emmaus Medical, Inc. (Industry)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10478; NCT00029887 (obsolete NCT alias)
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Results first posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2020-12

CONDITIONS: Sickle Cell Anemia; Thalassemia
Keywords: sickle cell disease; sickle cell anemia; L-glutamine; Sickle Cell Anemia (homozygous); Sickle ß0-Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia | interventions — Glutamine; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- investigational product (Experimental): L-glutamine
  Interventions: Drug: L-glutamine
- placebo (Placebo Comparator): maltodextrin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-glutamine — Approximately 0.3 g/kg total daily dose of L-glutamine will be orally administered (over two doses), with a maximum total daily dose of 30 grams.
  Other Names: oral L-glutamine
  Arms: investigational product
Drug: Placebo — Approximately 0.3 g/kg total daily dose of maltodextrin placebo will be orally administered (over two doses), with a maximum total daily dose of 30 grams.
  Other Names: maltodextrin
  Arms: placebo

SUMMARY:
The purpose of this research is to evaluate the effects of L-glutamine as a therapy for sickle cell anemia and sickle ß0-thalassemia. as evaluated by the number of occurrences of sickle cell crises.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the effectiveness of oral L-glutamine in the therapy of sickle cell anemia and sickle ß0-thalassemia.

The secondary purpose is to assess the effect of L-glutamine frequency of hospitalizations for sickle cell pain, frequency of emergency room visits for sickle cell pain; energy and appetite levels; narcotics usage.

Methodology:

By site, patients will be randomized to L-glutamine or placebo in a 1:1 ratio after a 4-week screening period. Patients will undergo 48 weeks of treatment with dosing BID orally, with dose calculated according to patient weight. Patient visits will occur every 4 weeks. After 48 weeks of treatment, dose will be tapered to zero within 3 weeks. A final evaluation visit will occur 2 weeks after last dose.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in the study, a patient must meet all of the following inclusion criteria:

* Patient is at least five years of age.
* Patient has been diagnosed with sickle cell anemia or sickle ß0-thalassemia (documented by hemoglobin electrophoresis).
* Patient has had at least two episodes of painful crises within 12 months of the screening visit.
* If the patient has been treated with an anti-sickling agent within three months of the screening visit, the therapy must have been continuous for at least three months with the intent to continue for the next 14 months.
* Patient or the patient's legally authorized representative has given written informed consent.
* If the patient is a female of child-bearing potential, she agrees to practice a recognized form of birth control during the course of the study.

Exclusion Criteria:

If the patient meets any of the following criteria, the patient must not be enrolled:

* Patient has a significant medical condition that required hospitalization (other than sickle painful crisis) within two months of the screening visit.
* Patient has diabetes mellitus with untreated fasting blood sugar >115 mg/dL.
* Patient has prothrombin time International Normalized Ratio (INR) > 2.0.
* Patient has serum albumin < 3.0 g/dl.
* Patient has received any blood products within three weeks of the screening visit.
* Patient has a history of uncontrolled liver disease or renal insufficiency.
* Patient is pregnant or lactating.
* Patient has been treated with an experimental anti-sickling medication/treatment (except hydroxyurea) within 30 days of the screening visit.
* Patient has been treated with an experimental drug within 30 days of the screening visit.
* There are factors that would, in the judgment of the investigator, make it difficult for the patient to comply with the requirements of the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2004-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka Niihara, MD, Principal Investigator — CEO, Emmaus Medical, Inc
Locations (5):
- United States (5):
  - Kaiser Permanente, Bellflower, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Grady Memorial Hospital, Atlanta, Georgia
  - University of Medicine and Dentistry, New Jersey, New Brunswick, New Jersey
  - Jacobi Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bolarinwa AB, Oduwole O, Okebe J, Ogbenna AA, Otokiti OE, Olatinwo AT. Antioxidant supplementation for sickle cell disease. Cochrane Database Syst Rev. 2024 May 22;5(5):CD013590. doi: 10.1002/14651858.CD013590.pub2. PMID 38775255

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Product | Placebo
Started | 37 | 33
Completed | 33 | 29
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: The full analysis dataset included all patients who received at least one dose of study medication and had been diagnosed with sickle cell anemia or sickle β°-thalassemia documented by hemoglobin electrophoresis and had at least 2 episodes of painful crises within 12 months prior to the screening visit (N = 62).
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Product | Placebo | Total
Number analyzed (Participants) | 33 | 29 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 6
  Between 18 and 65 years | 30 | 26 | 56
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (10.09) | 26.5 (9.42) | 28.6 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 10 | 32
  Male | 11 | 19 | 30
Region of Enrollment [Number; unit: participants]
  United States | 33 | 29 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Occurrences of Painful Sickle Cell Crises
Description: The mean number of painful sickle crisis through week 48
Time Frame: From Week 0 through Week 48 (cumulative)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Crisis
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
Crisis | 4.5 (5.37) | 10.8 (18.74)
Statistical Analysis 1: Comparison: Investigational Product vs Placebo; Test type: Superiority; p = 0.076, Cochran-Mantel-Haenszel

2. Secondary Outcome: Frequency of Hospitalizations for Sickle Cell Pain
Description: The mean number of hospitalizations through week 48
Time Frame: From Week 0 through Week 48 (cumulative)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Hosptalizations
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
Hosptalizations | 1.5 (2.46) | 2.3 (2.42)
Statistical Analysis 1: Comparison: Investigational Product vs Placebo; Test type: Superiority; p = 0.072, Cochran-Mantel-Haenszel

3. Secondary Outcome: Frequency of Emergency Room Visits for Sickle Cell Pain
Description: The mean number of emergency room visits through week 48
Time Frame: From Week 0 through Week 48 (cumulative)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Emergency room visits
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
Emergency room visits | 3.7 (5.63) | 9.4 (19.91)
Statistical Analysis 1: Comparison: Investigational Product vs Placebo; Test type: Superiority; p = 0.129, Cochran-Mantel-Haenszel

4. Secondary Outcome: The Effect of Oral L-glutamine on Hematological Parameters - Hemoglobin
Description: Patient's hemoglobin will be collected at each visit.Change from Baseline will be reported at Weeks 4, 24 and 40.
Time Frame: Baseline, Weeks 4, 24 and 40
Population: The safety population included all patients who received at least one dose of study medication (N = 70).
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 37 | 33
g/dL
  Baseline | 8.96 (1.477) | 9.05 (1.219)
  Change in Hemoglobin at Week 4: number analyzed (Participants) | 34 | 27
  Change in Hemoglobin at Week 4 | 0.15 (0.831) | -0.13 (0.861)
  Change in Hemoglobin at Week 24: number analyzed (Participants) | 22 | 21
  Change in Hemoglobin at Week 24 | 0.26 (0.641) | 0.16 (0.607)
  Change in Hemoglobin at Week 40: number analyzed (Participants) | 18 | 12
  Change in Hemoglobin at Week 40 | 0.11 (0.749) | -0.07 (0.650)

5. Secondary Outcome: The Effect of Oral L-glutamine on Hematological Parameters - Hematocrit
Description: Patient's hematocrit will be collected at each visit. Change from Baseline will be reported at Weeks 4, 24 and 40
Time Frame: Baseline, Weeks 4, 24, and 40
Population: The safety population included all patients who received at least one dose of study medication (N = 70).
Measure: Mean (Standard Deviation); unit: % RBC
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 37 | 33
% RBC
  Baseline | 25.90 (4.493) | 26.22 (4.125)
  Change in Hematocrit at Week 4: number analyzed (Participants) | 34 | 27
  Change in Hematocrit at Week 4 | 0.51 (2.784) | -0.09 (2.279)
  Change in Hematocrit at Week 24: number analyzed (Participants) | 22 | 21
  Change in Hematocrit at Week 24 | 1.08 (2.352) | 0.58 (2.050)
  Change in Hematocrit at Week 40: number analyzed (Participants) | 18 | 12
  Change in Hematocrit at Week 40 | 0.49 (2.786) | 0.26 (1.869)

6. Secondary Outcome: The Effect of Oral L-glutamine on Hematological Parameters - Reticulocyte Count
Description: Patient's reticulocyte count will be collected at each visit. Change from Baseline will be reported at Weeks 4, 24 and 40
Time Frame: Baseline, Weeks 0, 4, 24, 40
Population: The safety population included all patients who received at least one dose of study medication (N = 70).
Measure: Mean (Standard Deviation); unit: 10^12 Reticulocytes/L
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 37 | 33
10^12 Reticulocytes/L
  Baseline | 0.266 (0.1125) | 0.295 (0.0979)
  Change in Reticulocyte count at Week 4: number analyzed (Participants) | 19 | 14
  Change in Reticulocyte count at Week 4 | -0.040 (0.0993) | -0.034 (0.0689)
  Change in Reticulocyte count at Week 24: number analyzed (Participants) | 12 | 8
  Change in Reticulocyte count at Week 24 | -0.022 (0.0917) | -0.032 (0.1032)
  Change in Reticulocyte count at Week 40: number analyzed (Participants) | 10 | 3
  Change in Reticulocyte count at Week 40 | -0.016 (0.1357) | -0.020 (0.0908)

7. Secondary Outcome: Number of Participants With Narcotic Usage
Description: Analysis of narcotic usage was performed for the subset of patients with any narcotic use who completed the study. Changes in narcotic usage were determined by an independent consultant prior to database lock using morphine equivalents to determine relative use.
Time Frame: Week 24, Week 48
Population: Patients with any narcotic use who completed the visit
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 17 | 16
Participants
  Change in Narcotic Usage at Week 24: Change to weaker narcotics | 6 | 2
  Change in Narcotic Usage at Week 24: No change | 10 | 9
  Change in Narcotic Usage at Week 24: Change to stronger narcotics | 1 | 5
  Change in Narcotic Usage at Week 48: Change to weaker narcotics | 6 | 2
  Change in Narcotic Usage at Week 48: No change | 10 | 9
  Change in Narcotic Usage at Week 48: Change to stronger narcotics | 1 | 5

8. Secondary Outcome: Energy Level (11-point Scale)
Description: The patient's energy level was evaluated at each visit using an 11 point scale from 0=extremely tired to 10=extremely energetic
Time Frame: Collected at Week 0, 8, 16, 24, 32, 40, 48
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
score on a scale
  Week 0 | 6.1 (1.92) | 6.8 (1.99)
  Week 8: number analyzed (Participants) | 26 | 21
  Week 8 | 6.9 (1.84) | 7.1 (1.96)
  Week 16: number analyzed (Participants) | 28 | 21
  Week 16 | 6.9 (2.02) | 7.1 (2.70)
  Week 24: number analyzed (Participants) | 21 | 18
  Week 24 | 7.3 (1.65) | 7.8 (2.02)
  Week 32: number analyzed (Participants) | 19 | 14
  Week 32 | 7.3 (1.67) | 7.4 (1.95)
  Week40: number analyzed (Participants) | 18 | 13
  Week40 | 6.6 (1.54) | 6.9 (2.29)
  Week 48: number analyzed (Participants) | 24 | 22
  Week 48 | 6.8 (1.92) | 7.3 (1.83)

9. Secondary Outcome: Patient Appetite (3-point Scale)
Description: Patient's appetite level was evaluated at each visit using a 3 point scale: above average, average and below average. The parentages of patient at each visit whose appetite level was below, normal or above average were compared using CMH test (row mean scores) controlling for study center.
Time Frame: Collected at Week 0, 8, 16, 24, 32, 40, 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
Participants
  Patient appetite since the last visit - Visit 0: Above average | 4 | 6
  Patient appetite since the last visit - Visit 0: Average | 24 | 22
  Patient appetite since the last visit - Visit 0: Below average | 5 | 1
  Patient appetite since the last visit - Visit 0: Not known | 0 | 0
  Patient appetite since the last visit - Visit 8: number analyzed (Participants) | 26 | 22
  Patient appetite since the last visit - Visit 8: Above average | 4 | 6
  Patient appetite since the last visit - Visit 8: Average | 19 | 14
  Patient appetite since the last visit - Visit 8: Below average | 2 | 2
  Patient appetite since the last visit - Visit 8: Not known | 1 | 0
  Patient appetite since the last visit - Visit 16: number analyzed (Participants) | 28 | 22
  Patient appetite since the last visit - Visit 16: Above average | 3 | 9
  Patient appetite since the last visit - Visit 16: Average | 18 | 11
  Patient appetite since the last visit - Visit 16: Below average | 7 | 2
  Patient appetite since the last visit - Visit 16: Not known | 0 | 0
  Patient appetite since the last visit - Visit 24: number analyzed (Participants) | 22 | 20
  Patient appetite since the last visit - Visit 24: Above average | 4 | 7
  Patient appetite since the last visit - Visit 24: Average | 17 | 11
  Patient appetite since the last visit - Visit 24: Below average | 1 | 2
  Patient appetite since the last visit - Visit 24: Not known | 0 | 0
  Patient appetite since the last visit - Visit 32: number analyzed (Participants) | 19 | 15
  Patient appetite since the last visit - Visit 32: Above average | 3 | 3
  Patient appetite since the last visit - Visit 32: Average | 15 | 12
  Patient appetite since the last visit - Visit 32: Below average | 1 | 0
  Patient appetite since the last visit - Visit 32: Not known | 0 | 0
  Patient appetite since the last visit - Visit 40: number analyzed (Participants) | 18 | 13
  Patient appetite since the last visit - Visit 40: Above average | 2 | 4
  Patient appetite since the last visit - Visit 40: Average | 13 | 7
  Patient appetite since the last visit - Visit 40: Below average | 3 | 2
  Patient appetite since the last visit - Visit 40: Not known | 0 | 0
  Patient appetite since the last visit - Visit 48: number analyzed (Participants) | 17 | 12
  Patient appetite since the last visit - Visit 48: Above average | 2 | 2
  Patient appetite since the last visit - Visit 48: Average | 13 | 9
  Patient appetite since the last visit - Visit 48: Below average | 2 | 1
  Patient appetite since the last visit - Visit 48: Not known | 0 | 0

10. Secondary Outcome: The Effect of Oral L-glutamine on Vital Signs - Blood Pressure
Description: Patient's blood pressure will be collected at each visit. Change from Baseline will be reported at Weeks 4, 24, and 48
Time Frame: Baseline, Weeks 4, 24, and 48
Population: The safety population included all patients who received at least one dose of study medication (N = 70).
Measure: Mean (Standard Deviation); unit: mm/Hg
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 37 | 33
mm/Hg
  Baseline SBP (mm/Hg) | 115.18 (14.30) | 119.6 (13.64)
  Change in SBP (mm/Hg) at Week 4: number analyzed (Participants) | 33 | 26
  Change in SBP (mm/Hg) at Week 4 | 0.7 (10.98) | -0.9 (10.81)
  Change in SBP (mm/Hg) at Week 24: number analyzed (Participants) | 23 | 20
  Change in SBP (mm/Hg) at Week 24 | 2.2 (10.48) | -1.9 (13.06)
  Change in SBP (mm/Hg) at Week 48: number analyzed (Participants) | 18 | 13
  Change in SBP (mm/Hg) at Week 48 | -1.2 (12.07) | -1.5 (12.97)
  Baseline DBP (mm/hg) | 63.7 (9.05) | 64.9 (8.09)
  Change in DBP (mm/Hg) at Week 4: number analyzed (Participants) | 33 | 26
  Change in DBP (mm/Hg) at Week 4 | 1.2 (8.09) | 2.2 (8.73)
  Change in DBP (mm/Hg) at Week 24: number analyzed (Participants) | 23 | 20
  Change in DBP (mm/Hg) at Week 24 | 1.2 (9.55) | -0.4 (6.88)
  Change in DBP (mm/Hg) at Week 48: number analyzed (Participants) | 18 | 13
  Change in DBP (mm/Hg) at Week 48 | -1.3 (7.98) | 0.5 (7.91)

11. Secondary Outcome: The Effect of Oral L-glutamine on Vital Signs - Temperature
Description: Patient's temperature will be collected at each visit. Change from Baseline will be reported at Weeks 4, 24, and 48
Time Frame: Baseline, Weeks 4, 24, and 48
Population: The safety population included all patients who received at least one dose of study medication (N = 70).
Measure: Mean (Standard Deviation); unit: deg C
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 37 | 33
deg C
  Baseline | 36.40 (0.686) | 36.29 (0.613)
  Change in Temperature at Week 4: number analyzed (Participants) | 33 | 27
  Change in Temperature at Week 4 | -0.05 (0.377) | -0.06 (0.269)
  Change Temperature at Week 24: number analyzed (Participants) | 23 | 20
  Change Temperature at Week 24 | -0.01 (0.261) | -0.07 (0.268)
  Change in Temperature at Week 48: number analyzed (Participants) | 18 | 13
  Change in Temperature at Week 48 | 0.08 (0.362) | -0.09 (0.256)

12. Secondary Outcome: The Effect of Oral L-glutamine on Vital Signs - Respiration
Description: Respiration will be collected at each visit. Change from Baseline will be reported at Weeks 4, 24, and 48
Time Frame: Baseline, Weeks 4, 24, and 48
Population: The safety population included all patients who received at least one dose of study medication (N = 70).
Measure: Mean (Standard Deviation); unit: resp/min
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 37 | 33
resp/min
  Baseline | 17.9 (2.11) | 17.7 (1.94)
  Change in Respiration at Week 4: number analyzed (Participants) | 33 | 27
  Change in Respiration at Week 4 | 0.3 (1.71) | 0.6 (1.58)
  Change in Respiration at Week 24: number analyzed (Participants) | 23 | 20
  Change in Respiration at Week 24 | 0.4 (1.73) | -0.4 (1.93)
  Change in Respiration at Week 48: number analyzed (Participants) | 18 | 13
  Change in Respiration at Week 48 | 0.4 (2.12) | 0.6 (2.47)

13. Secondary Outcome: The Effect of Oral L-glutamine on Vital Signs - Pulse Rate
Description: Patient's pulse rate will be collected at each visit, Change from Baseline will be reported at Weeks 4, 24, and 48
Time Frame: Baseline, Weeks 4, 24, and 48
Population: The safety population included all patients who received at least one dose of study medication (N = 70).
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 37 | 33
bpm
  Baseline | 81.6 (11.37) | 80.5 (11.95)
  Change in Pulse Rate at Week 4: number analyzed (Participants) | 33 | 27
  Change in Pulse Rate at Week 4 | 2.5 (12.88) | 0.7 (12.11)
  Change in Pulse Rate at Week 24: number analyzed (Participants) | 23 | 20
  Change in Pulse Rate at Week 24 | 1.7 (13.69) | -2.7 (12.81)
  Change in Pulse Rate at Week 48: number analyzed (Participants) | 18 | 13
  Change in Pulse Rate at Week 48 | 1.3 (14.53) | 3.9 (10.07)

14. Secondary Outcome: Effect of L-glutamine on Alcohol Use
Description: The patient's alcohol usage will be assessed at each visit. Alcohol usage will be reported at Weeks 0, 8,16, 24, 32, 40 and 48
Time Frame: Weeks 0, 8,16, 24, 32, 40 and 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
Participants
  Week 0: NO - Alcohol Use | 30 | 27
  Week 0: YES - Alcohol Use | 3 | 2
  Week 8: number analyzed (Participants) | 26 | 22
  Week 8: NO - Alcohol Use | 25 | 20
  Week 8: YES - Alcohol Use | 1 | 2
  Week 16: number analyzed (Participants) | 28 | 22
  Week 16: NO - Alcohol Use | 27 | 20
  Week 16: YES - Alcohol Use | 1 | 2
  Week 24: number analyzed (Participants) | 22 | 20
  Week 24: NO - Alcohol Use | 22 | 19
  Week 24: YES - Alcohol Use | 0 | 1
  Week 32: number analyzed (Participants) | 19 | 15
  Week 32: NO - Alcohol Use | 19 | 13
  Week 32: YES - Alcohol Use | 0 | 2
  Week 40: number analyzed (Participants) | 18 | 13
  Week 40: NO - Alcohol Use | 18 | 11
  Week 40: YES - Alcohol Use | 0 | 2
  Week 48: number analyzed (Participants) | 17 | 12
  Week 48: NO - Alcohol Use | 17 | 11
  Week 48: YES - Alcohol Use | 0 | 1

15. Secondary Outcome: Effect of L-glutamine on Tobacco Use
Description: Patient's alcohol usage will be assessed at each visit. Alcohol usage will be reported at Weeks 0, 8,16, 24, 32, 40 and 48
Time Frame: Weeks 0, 8,16, 24, 32, 40 and 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
Participants
  Week 0: NO - Tobacco use | 28 | 27
  Week 0: YES - Tobacco use | 5 | 2
  Week 8: number analyzed (Participants) | 26 | 22
  Week 8: NO - Tobacco use | 23 | 21
  Week 8: YES - Tobacco use | 3 | 1
  Week 16: number analyzed (Participants) | 28 | 22
  Week 16: NO - Tobacco use | 24 | 22
  Week 16: YES - Tobacco use | 4 | 0
  Week 24: number analyzed (Participants) | 22 | 20
  Week 24: NO - Tobacco use | 20 | 19
  Week 24: YES - Tobacco use | 2 | 1
  Week 32: number analyzed (Participants) | 19 | 15
  Week 32: NO - Tobacco use | 18 | 15
  Week 32: YES - Tobacco use | 1 | 0
  Week 40: number analyzed (Participants) | 18 | 13
  Week 40: NO - Tobacco use | 17 | 13
  Week 40: YES - Tobacco use | 1 | 0
  Week 48: number analyzed (Participants) | 17 | 12
  Week 48: NO - Tobacco use | 16 | 12
  Week 48: YES - Tobacco use | 1 | 0

16. Secondary Outcome: The Effect of Oral L-glutamine on the Number of Days Patient's Daily Activities Are Interrupted Due to Sickle Cell Pain
Description: Percentage of days a patient's daily activities were interrupted due to sickle pain calculated at each visit. Day's interrupted will be reported at Weeks 0, 8,16, 24, 32, 40 and 48
Time Frame: Weeks 0, 8,16, 24, 32, 40 and 48
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: % of days interrupted
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
% of days interrupted
  Week 0 | 8.3 (11.19) | 8.1 (11.94)
  Week 8: number analyzed (Participants) | 25 | 22
  Week 8 | 11.9 (21.22) | 24.2 (29.22)
  Week 16: number analyzed (Participants) | 28 | 22
  Week 16 | 23.3 (28.56) | 15.5 (21.55)
  Week 24: number analyzed (Participants) | 22 | 19
  Week 24 | 11.4 (18.34) | 11.7 (12.75)
  Week 32: number analyzed (Participants) | 19 | 15
  Week 32 | 12.5 (17.96) | 15.7 (17.33)
  Week 40: number analyzed (Participants) | 18 | 13
  Week 40 | 13.2 (16.88) | 28.0 (31.33)
  Week 48: number analyzed (Participants) | 17 | 11
  Week 48 | 11.7 (19.17) | 11.5 (17.58)

17. Secondary Outcome: The Effect of Oral L-glutamine on Subjective Quality of Life
Description: The subjective quality of life was evaluated using the scoring of the RAND 36-Item Health Survey Questionnaire. The subjective quality of life (Physical functioning, Physical health, Emotional problems, Energy/Fatigue, Emotional well being, Social functioning, Pain, General health) will be reported at Baseline and Week 24 (or at time of discontinuation). The range for Physical functioning, Physical health, Emotional problems, Emotional well being and Social functioning is 0-100, with a high score denotes a better quality of life. For Energy/Fatigue, Pain and General health the range is 0-100, with a lower score denotes better quality of life.
Time Frame: Baseline and Week 24 (or at time of discontinuation)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
score on a scale
  Physical Functioning Baseline: number analyzed (Participants) | 31 | 27
  Physical Functioning Baseline | 61.7 (25.38) | 69.9 (26.68)
  Physical Functioning Week 24: number analyzed (Participants) | 28 | 25
  Physical Functioning Week 24 | 65.5 (23.18) | 76.0 (17.38)
  Physical Health - Baseline: number analyzed (Participants) | 31 | 27
  Physical Health - Baseline | 43.5 (38.17) | 49.1 (40.72)
  Physical Health - Week 24: number analyzed (Participants) | 28 | 25
  Physical Health - Week 24 | 55.6 (41.79) | 46.7 (40.83)
  Emotional Problems - Baseline: number analyzed (Participants) | 31 | 27
  Emotional Problems - Baseline | 52.7 (41.97) | 66.7 (41.35)
  Emotional Problems - Week 24: number analyzed (Participants) | 28 | 25
  Emotional Problems - Week 24 | 58.3 (40.20) | 65.3 (40.24)
  Energy/Fatigue - Baseline: number analyzed (Participants) | 31 | 27
  Energy/Fatigue - Baseline | 45.7 (12.29) | 50.0 (17.82)
  Energy/Fatigue - Week 24: number analyzed (Participants) | 28 | 25
  Energy/Fatigue - Week 24 | 49.8 (19.65) | 53.4 (21.96)
  Emotional Well Being - Baseline: number analyzed (Participants) | 31 | 27
  Emotional Well Being - Baseline | 66.2 (19.37) | 74.5 (16.02)
  Emotional Well Being - Week 24: number analyzed (Participants) | 28 | 25
  Emotional Well Being - Week 24 | 71.9 (17.83) | 77.1 (21.92)
  Social Functioning - Baseline: number analyzed (Participants) | 31 | 27
  Social Functioning - Baseline | 61.3 (24.01) | 62.5 (24.27)
  Social Functioning - Week 24: number analyzed (Participants) | 20 | 16
  Social Functioning - Week 24 | 72.5 (22.06) | 65.6 (26.02)
  Pain - Baseline: number analyzed (Participants) | 31 | 27
  Pain - Baseline | 53.4 (23.41) | 55.5 (28.07)
  Pain - Week 24: number analyzed (Participants) | 28 | 25
  Pain - Week 24 | 59.1 (24.60) | 56.1 (30.76)
  General Health - Baseline: number analyzed (Participants) | 31 | 27
  General Health - Baseline | 46.0 (17.42) | 49.7 (21.5)
  General Health - Week 24: number analyzed (Participants) | 28 | 25
  General Health - Week 24 | 53.9 (16.55) | 57.0 (18.62)

18. Secondary Outcome: Effect of Oral L--glutamine on Height
Description: Height will be measured at each visit. Change from Baseline will be reported at Weeks 4, 24, and 48
Time Frame: Baseline, Weeks 4, 24, and 48
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
cm
  Baseline | 169.8 (9.49) | 169.2 (11.87)
  Change in Height at Week 4: number analyzed (Participants) | 31 | 24
  Change in Height at Week 4 | -0.1 (1.18) | 0.2 (2.87)
  Change in Height at Week 24: number analyzed (Participants) | 22 | 19
  Change in Height at Week 24 | 0.1 (1.54) | -0.1 (1.68)
  Change in Height at Week 48: number analyzed (Participants) | 17 | 12
  Change in Height at Week 48 | -1.7 (6.58) | 0.4 (3.35)

19. Secondary Outcome: Effect of Oral L--glutamine on Weight
Description: Weight will be measured at each visit. Change from Baseline will be reported at Weeks 4, 24, and 48
Time Frame: Baseline, Weeks 4, 24 and 48
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
kg
  Baseline | 67.1 (13.39) | 70.7 (18.20)
  Change in Weight at Week 4: number analyzed (Participants) | 31 | 24
  Change in Weight at Week 4 | 0.8 (1.89) | 0.1 (3.13)
  Change in Weight at Week 24: number analyzed (Participants) | 22 | 19
  Change in Weight at Week 24 | 1.2 (2.55) | 1.4 (5.04)
  Change in Weight at Week 48: number analyzed (Participants) | 17 | 12
  Change in Weight at Week 48 | -1.0 (10.79) | 1.9 (7.39)

20. Secondary Outcome: Effect of L-glutamine on Subjective Exercise Tolerance - Minutes Patient Could Walk Without Rest
Description: Minutes patient could walk without rest will be measured at each visit. Change from Baseline will be reported at Weeks 4, 24, and 48.
Time Frame: Baseline, Weeks 4, 24, and 48.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mins
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
mins
  Baseline - Minutes patient could walk without rest | 32 (28.25) | 28.6 (23.94)
  Change in Minutes patient could walk without rest at Week 4: number analyzed (Participants) | 32 | 24
  Change in Minutes patient could walk without rest at Week 4 | -2.1 (29.57) | -1.8 (20.06)
  Change in Minutes patient could walk without rest at Week 24: number analyzed (Participants) | 22 | 20
  Change in Minutes patient could walk without rest at Week 24 | -1.9 (26.30) | -3.5 (12.63)
  Change in Minutes patient could walk without rest at Week 48: number analyzed (Participants) | 17 | 12
  Change in Minutes patient could walk without rest at Week 48 | -5.8 (24.88) | 6.7 (28.95)

21. Secondary Outcome: Effect of L-glutamine on Subjective Exercise Tolerance - Minutes Patient Could Run Without Rest
Description: Minutes patient could run without rest will be measured at each visit. Change from Baseline will be reported at Weeks 4, 24, and 48.
Time Frame: Baseline, Weeks 4, 24, and 48.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mins
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
mins
  Baseline - Minutes patient could run without rest | 5.1 (8.90) | 7.4 (10.02)
  Change in Minutes patient could run without rest at Week 4: number analyzed (Participants) | 32 | 24
  Change in Minutes patient could run without rest at Week 4 | -0.7 (4.75) | -0.7 (8.64)
  Change in Minutes patient could run without rest at Week 24: number analyzed (Participants) | 22 | 20
  Change in Minutes patient could run without rest at Week 24 | -0.3 (5.17) | -1.2 (13.56)
  Change in Minutes patient could run without rest at Week 48: number analyzed (Participants) | 17 | 12
  Change in Minutes patient could run without rest at Week 48 | -0.8 (5.14) | -1.2 (12.78)

22. Secondary Outcome: Effect of L-glutamine on Subjective Exercise Tolerance - Distance Patient Could Walk Without Rest
Description: Distance patient could walk without rest will be collected at each visit. Change from Baseline will be reported at Weeks 4, 24, and 48.
Time Frame: Baseline, Weeks 4, 24, and 48.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
feet
  Baseline - Distance patient could walk without rest | 4097.5 (2739) | 5680.7 (7695)
  Change in Distance patient could walk without rest at Week 4: number analyzed (Participants) | 32 | 24
  Change in Distance patient could walk without rest at Week 4 | 41.9 (1976) | 302.5 (2022)
  Change in Distance patient could walk without rest at Week 24: number analyzed (Participants) | 22 | 20
  Change in Distance patient could walk without rest at Week 24 | 74.5 (2116) | -1719 (9569)
  Change in Distance patient could walk without rest at Week 48: number analyzed (Participants) | 17 | 12
  Change in Distance patient could walk without rest at Week 48 | 38.8 (2766) | -4240 (11782)

23. Secondary Outcome: Effect of L-glutamine on Subjective Exercise Tolerance - Distance Patient Could Run Without Rest
Description: Distance patient could run without rest will be collected at each visit. Change from Baseline will be reported at Weeks 4, 24, and 48.
Time Frame: Baseline, Weeks 4, 24, and 48.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Investigational Product | Placebo
Number analyzed (Participants) | 33 | 29
feet
  Baseline - Distance patient could run without rest | 1059.5 (1688) | 1482.1 (2160)
  Change in Distance patient could run without rest at Week 4: number analyzed (Participants) | 32 | 24
  Change in Distance patient could run without rest at Week 4 | -31.6 (1054) | 124.2 (1226)
  Change in Distance patient could run without rest at Week 24: number analyzed (Participants) | 22 | 20
  Change in Distance patient could run without rest at Week 24 | 215.9 (1411) | 186.5 (2901)
  Change in Distance patient could run without rest at Week 48: number analyzed (Participants) | 17 | 12
  Change in Distance patient could run without rest at Week 48 | 13.5 (1677) | -586.7 (2698)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected throughout the course of the study (53 weeks or about 1 year).
Description: The Safety population will include all patients who received at least one dose of study medication.
Arm/Group | Investigational Product | Placebo
All-Cause Mortality (participants affected / at risk) | 1/37 | 0/33
Serious Adverse Events (participants affected / at risk) | 24/37 | 21/33
Other Adverse Events (participants affected / at risk) | 37/37 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Product (N=37) | Placebo (N=33)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 22 (22) | 17 (17)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
pyrexia (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
URTI (Infections and infestations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hip Arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Product (N=37) | Placebo (N=33)
Sickle cell anemia with crisis (Congenital, familial and genetic disorders) | 31 (31) | 26 (26)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Influenza-like illness (General disorders) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3)
Gastroenteritis (Infections and infestations) | 2 (2) | 5 (5)
URTI (Infections and infestations) | 1 (1) | 3 (3)
Ear infection (Infections and infestations) | 0 (0) | 2 (2)
Gastroentritis viral (Infections and infestations) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees that any INFORMATION submitted to it by EMMAUS shall be maintained in secrecy for a period of seven (7) years from each disclosure of INFORMATION. PI will use the up most due diligence to prevent disclosure by it except to its employees, agents, and contractors necessary for evaluation, all of whom shall be bound by similar written obligations of confidentiality, and who agree not to use the INFORMATION for any purpose other than for evaluation purposes.